CLINICAL TRIAL: NCT00619658
Title: The Feasibility of Simplified Telephone Follow-up After Medical Abortion
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO07080379
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Induced Abortion
Keywords: telephone follow-up; medical abortion; induced abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All women undergoing medical abortion will have telephone follow-up approximately one week after using mifepristone and misoprostol.
  Interventions: Other: telephone follow-up

INTERVENTIONS:
Other: telephone follow-up — subjects undergoing medical abortion will recieve a telephone call and be asked a series of clinical questions. Expulsion of the pregnancy will be assessed based on the answers to those questions.

SUMMARY:
To assess the feasibility of using simplified telephone follow-up to predict pregnancy expulsion after medical abortion, and if in-person follow-up is required to determine the percentage of women that will present for that follow-up.

DETAILED DESCRIPTION:
This is a prospective trial to evaluate the feasibility of performing a telephone interview to predict if pregnancy expulsion has occurred. In those women for whom expulsion has not been predicted to have occurred, the trial will evaluate if they will present for a follow-up visit. We plan to recruit 154 women that desire a medical abortion from Magee-Womens Hospital, Planned Parenthood of Western Pennsylvania, and private offices in the surrounding area. Women who are no more than 63 days gestation will receive mifepristone 200mg and misoprostol 800mcg. Each subject will choose between two evidence-based methods of using the misoprostol: buccally 24-72 hours or vaginally 0-72 hours after mifepristone. A follow-up phone call with a clinician will occur 5-9 days after mifepristone administration. Based on clinical history, including a structured question set, the subject and the clinician will predict if expulsion occurred. If either or both feel that expulsion may not have occurred, the women will return for follow-up in the office within one week for sonographic evaluation. If they both predict that expulsion has occurred at this initial phone call follow-up, the subject will perform a urine pregnancy test at home in approximately 3 weeks. She will have a follow-up phone call after the pregnancy test to obtain the results. The subject will only have an additional visit and ultrasound examination if the urine pregnancy test is positive.

The primary outcome is the percentage of women that will be available for follow-up over the phone, and/or return visit if necessary. The secondary outcomes are to determine if a standardized set of questions of clinical history after medical abortion will be useful to predict expulsion of the pregnancy and which mode of misoprostol administration women prefer. In addition, the study will confirm if women and clinicians are accurate at predicting expulsion of the pregnancy, compare the ability of patients and clinicians to predict expulsion of the pregnancy, determine how many women require follow-up evaluation after a telephone interview, and to determine the pregnancy continuation rate after misoprostol and mifepristone in this study.

ELIGIBILITY:
Inclusion Criteria:

* healthy females
* requesting an elective termination of pregnancy by medical abortion
* an intrauterine pregnancy </= 63 days gestation
* willing and able to sign the informed consent
* willing to comply with the study protocol and visit schedule
* willing to have a surgical abortion/D&C if indicated
* with easy and ready access to a telephone

Exclusion Criteria:

* contraindication to mifepristone
* contraindication to misoprostol
* cardiovascular disease -hemoglobin <10 g/dL
* known clotting defect or receiving anticoagulants
* pregnancy with an IUD
* breastfeeding
* ultrasound evidence of an early pregnancy failure
* pelvic examination with evidence of acute cervicitis
* prior participation in this research study
* current participation in a conflicting research study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine the rate of completion of telephone interviews after medical abortion, and the rate of return for follow-up if necessary. | four months

SECONDARY OUTCOMES:
To determine if a standardized set of questions can predict pregnancy expulsion, and to determine which method of misoprostol administration women prefer. | four months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Perriera, MD, Principal Investigator — Center for Family Planning Research, University of Pittsburgh
Locations (1):
- Center for Family Planning Research, Magee-Womens Hospital, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Rossi B, Creinin MD, Meyn LA. Ability of the clinician and patient to predict the outcome of mifepristone and misoprostol medical abortion. Contraception. 2004 Oct;70(4):313-7. doi: 10.1016/j.contraception.2004.04.005. PMID 15451336
- See also: Center for Family Planning Research website — http://www.birthcontrolstudies.org